CLINICAL TRIAL: NCT04828421
Title: The Effect of Probiotic Supplementation on Cognitive and Emotional Functions in Healthy Elderly Subjects: a Randomized, Double-blind, Cross-over and Controlled Trial
Brief Title: The Effect of Probiotic Supplementation on Cognitive and Emotional Functions in Healthy Elderly Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Almeria (Other)
Responsible Party: Principal Investigator, Pablo Román López, Principal Investigator, Vicedean of Nursing, Universidad de Almeria
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: UALBIO2020/001
Record Dates: First submitted 2021-03-29; First posted 2021-04-02 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Healthy
Keywords: Probiotics; Cognitive; Emotional; Aging; Elderly

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic group (Experimental): Participants will be treated with a daily capsule of a multi-species probiotic (3.3 billion Lactobacillus rhamnosus and Bifidobacterium lactis) during 10 weeks.
  Interventions: Dietary Supplement: Lactobacillus rhamnosus and Bifidobacterium lactis
- Placebo group (Placebo Comparator): Participants will receive a harmless substance (potato starch) during 10 weeks.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Lactobacillus rhamnosus and Bifidobacterium lactis — Probiotics
  Arms: Probiotic group
Dietary Supplement: Placebo — Placebo
  Arms: Placebo group

SUMMARY:
This study evaluates the cognitive and emotional effects of probiotics in healthy elderly patients.

DETAILED DESCRIPTION:
Gut microbiota (GM) has focused as an important target for emotional and cognitive diseases, moreover in a population that show an altered GM such as elderly population as age-related changes. Several studies have shown that ageing alter GM, both in diversity and integrity.

Probiotics have demonstrated that correct or prevent age-related dysbiosis, in order to reduce or prevent intestinal permeability and associated inflammation, inhibit the generation of harmful and/or toxic metabolites, as well as promote the production of beneficial bacterial components.

The aim of this study is to assess the effectiveness of a multiprobiotic formulation as a therapeutic strategy to attenuate the emotional and cognitive decline associated with ageing in healthy adults over 55 years of age. The hypothesis is that administration of a multi-species probiotic for 10 weeks will slow and/or ameliorate the decline in emotional and cognitive function inherent to senescence.

ELIGIBILITY:
Inclusion Criteria:

* be aged 55 years or over,
* voluntarily agree to participate in the study in accordance with the Helsinki declaration,
* not be participating in another study that could interfere with the results.

Exclusion Criteria:

* suffer from any serious mental illness other than depression and anxiety,
* score below 10 on the Mini-Mental State Examination (MMSE) (severe cognitive impairment)
* be using medications that affect cognition,
* taking anti-inflammatory drugs, antipsychotics, antibiotics and/or anxiolytics,
* have a serious illness (e.g. cancer, Parkinson's or Alzheimer's).

Min Age: 56 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2020-07-17 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Anxiety at 10 weeks | Before and after treatment (10 weeks)
  The State-Trait Anxiety Inventory. Score range: 20-80
Change from Baseline Depression at 10 weeks | Before and after treatment (10 weeks)
  The Beck Depression Inventory. Score range: 0-63.
Change from Baseline General Cognitive Status at 10 weeks | Before and after treatment (10 weeks)
  Mini-Mental State Examination. Score range: 0-35
Change from Baseline Working Memory at 10 weeks | Before and after treatment (10 weeks)
  Digits task, Corsi task
Change from Baseline Planning Ability at 10 weeks | Before and after treatment (10 weeks)
  Tower of London test
Change from Baseline Problem-solving ability at 10 weeks | Before and after treatment (10 weeks)
  Wisconsin Card Sorting test
Change from Baseline Selective attention, cognitive flexibility and response inhibition at 10 weeks | Before and after treatment (10 weeks)
  Stroop task
Change from Baseline Visual Attention at 10 weeks | Before and after treatment (10 weeks)
  Trail Making Test
Change from Baseline Motor impulsivity or inhibitory response at 10 weeks | Before and after treatment (10 weeks)
  Go/No-Go task
Change from Baseline Choice impulsivity or impulsive decision-making at 10 weeks | Before and after treatment (10 weeks)
  Iowa Gambling Task

SECONDARY OUTCOMES:
Change from Baseline Food Habits at 10 weeks | Before and after treatment (10 weeks)
  "24-hour recall" questionnaire
Change from Baseline Alcohol Use at 10 weeks | Before and after treatment (10 weeks)
  The Alcohol Use Disorders Identification Test. Score range: 0-40
Change from Baseline Body Composition at 10 weeks | Before and after treatment (10 weeks)
  Fat mass. Body fat mass. Fat-free mass. Total body water.
Change from Baseline Physical Activity at 10 weeks | Before and after treatment (10 weeks)
  International Physical Activity Questionnaire
Change from Baseline Stool Consistency at 10 weeks | Before and after treatment (10 weeks)
  The Bristol Scale
Change from Baseline Sleep Quality at 10 weeks | Before and after treatment (10 weeks)
  The Pittsburgh Sleep Quality Index Questionnaire. Score range: 0-21
Change from Baseline Perceived Stress at 10 weeks | Before and after treatment (10 weeks)
  Perceived Stress Questionnaire. Score range: 0-1
Change from Baseline Gastrointestinal Symptom at 10 weeks | Before and after treatment (10 weeks)
  Gastrointestinal Symptom Rating Scale

CONTACTS AND LOCATIONS:
Overall Officials: PABLO R LOPEZ, Principal Investigator — Universidad de Almeria
Locations (3):
- Spain (3):
  - Universidad de Almeria, Almería, Almeria
  - Universidad de Almeria, La Cañada de San Urbano, Almeria
  - Pablo Roman, Almería

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ruiz-Gonzalez C, Cardona D, Rueda-Ruzafa L, Rodriguez-Arrastia M, Ropero-Padilla C, Roman P. Cognitive and Emotional Effect of a Multi-species Probiotic Containing Lactobacillus rhamnosus and Bifidobacterium lactis in Healthy Older Adults: A Double-Blind Randomized Placebo-Controlled Crossover Trial. Probiotics Antimicrob Proteins. 2025 Oct;17(5):3525-3537. doi: 10.1007/s12602-024-10315-2. Epub 2024 Jun 27. PMID 38935259